CLINICAL TRIAL: NCT03720431
Title: A Phase 1b, Open-Label, Safety and Tolerability Study of TTAC-0001 in Combination With Pembrolizumab in Patients With Metastatic Triple-Negative Breast Cancer
Brief Title: TTAC-0001 and Pembrolizumab Phase Ib Combination Trial in Metastatic Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PharmAbcine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PMC_TTAC-0001_05
Record Dates: First submitted 2018-10-22; First posted 2018-10-25 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — olinvacimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TTAC-0001 and pembrolizumab (Experimental): TTAC-0001 and pembrolizumab combination therapy will be administered.
  Interventions: Drug: TTAC-0001 and pembrolizumab combination

INTERVENTIONS:
Drug: TTAC-0001 and pembrolizumab combination — * Investigational product (IP): TTAC-0001 and Pembrolizumab (Merck, Keytruda®)
  * Treatment groups: 3 dose levels
    * Dose level 1 (optimal starting dose): TTAC-0001 12 mg/kg on D1, D8 and D15 + Pembrolizumab 200 mg on D1
    * Dose level 2 (first escalation dose): TTAC-0001 16 mg/kg on D1, D8 and D15 + Pembrolizumab 200 mg on D1
    * Dose level 0 (de-escalation dose): TTAC-0001 8 mg/kg on D1, D8 and D15 + Pembrolizumab 200 mg on D1
  * Cycle: 3 weeks (21 days per cycle)

SUMMARY:
This is a phase 1b, open-Label clinical trial to determine the safety and tolerability and to establish a preliminary recommended Phase 2 dose (RP2D) of TTAC-0001 administered in combination with pembrolizumab in patients with metastatic triple-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients ≥18 years old
2. Histologically proven metastatic breast carcinoma with triple negative receptor status (Estrogen receptor, Progesterone receptor and human epidermal growth factor receptor 2 [HER2] negative) by IHC and Fluorescence in situ hybridization (FISH) according to ASCO-CAP guideline3.
3. At least one confirmed measurable lesion by RECIST 1.1 criteria
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
5. A person who satisfies the following criteria in hematologic, renal, and hepatic function tests performed within 7 days prior to screening:

(1) Hematologic tests

* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelets ≥ 100 x 109/L
* Haemoglobin ≥ 9.0 g/dL (2) Blood coagulation tests
* Prothrombin time (PT) ≤ 1.5 x Upper limit of normal (UNL)
* Activated partial thromboplastin Time (aPTT) ≤ 1.5 x UNL (3) Hepatic function tests
* Total bilirubin ≤ 1.5 x UNL
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 x ULN (≤ 5 x ULN in case of liver metastasis) (4) Renal function test
* ≤1.5 × ULN or creatinine clearance (CrCl) ≥30 mL/min for patient with creatinine levels >1.5 × institutional ULN 6) At least 12 weeks of expected life expectancy 7) The patient (or legally acceptable representative if applicable) is able and willing to provide written informed consent for the trial.

Exclusion Criteria:

1. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. (Note: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) controlled by curative therapy are not excluded)
2. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment
3. Has a history of (non-infectious) pneumonitis/interstitial lung diseases that required steroids or current pneumonitis/interstitial lung disease.
4. Has an active infection requiring systemic therapy
5. Uncontrolled hypertension (systolic blood pressure [SBP]> 150 or diastolic blood pressure [DBP]> 90 mmHg)
6. Uncontrolled seizures
7. Class III or IV heart failure by New York Heart Association (NYHA) classification
8. Has oxygen-dependent chronic disease
9. Active psychiatric disorder (schizophrenia, major depressive disorder, bipolar disorder etc.). Treated depression with ongoing antidepressant medication is not an exclusion
10. History of abdominal fistula or gastrointestinal perforation within 6 months prior to start of study drug
11. History of serious gastrointestinal haemorrhage within 6 months prior to start of study drug
12. History of severe arterial thromboembolic event within 12 months of start of study drug
13. Serious grade 4 venous thromboembolic event including pulmonary embolism
14. History of hypertensive crisis or hypertensive encephalopathy
15. History of posterior reversible encephalopathy syndrome
16. Planned surgery within 4 weeks post last dose
17. Moderate to severe proteinuria
18. Requiring therapeutic anticoagulation with warfarin at baseline
19. Not recovered below National Cancer Institute -Common Terminology Criteria for Adverse Events (NCI-CTCAE) grade 1 or baseline from AEs due to previous therapy
20. Treatment with systemic chemotherapy, hormonal therapy, immunotherapy or biologic therapy within 2 weeks prior to the baseline visit
21. Has received prior radiotherapy within 2 weeks of start of study treatment.
22. Undergone major surgery requiring general anaesthesia or a respiratory assistance device within 4 weeks prior to the baseline visit
23. Treated with other investigational drugs within 4 weeks prior to the baseline visit for this study
24. Female who is pregnant* or lactating and of childbearing potential who does not agree to a reliable and adequate method of contraception
25. A known history of severe drug hypersensitivity or hypersensitivity to a therapy similar to the study drugs
26. Unable to participate in the trial according to the investigator's decision.
27. Previous therapy with vascular endothelial growth factor (VEGF)-targeted agents including (but not limited to) bevacizumab
28. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) and was discontinued from that treatment due to a Grade 3 or higher irAE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2022-10-26 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities | During the first cycle (every cycle is 21 days) of treatment
  The frequency and percentage of DLT will be presented by dose level
Adverse events | From date of screening visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  The frequency and percentage of AEs will be presented by dose level
Immunogenicity | From date of screening visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Presence anti-drug antibody (ADA) will be listed

SECONDARY OUTCOMES:
Overall response rate | At every 2nd cycles until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years (every cycle is 21 days)]
  complete response (CR) or partial response (PR) by RECIST criteria
Disease control rate | At every 2nd cycles until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years (every cycle is 21 days)
  complete response (CR), partial response (PR) or stable disease (SD) by RECIST criteria
Progression free survival | From date of screening visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Period from the date of the drug administration to the disease progression time point
Overall survival | From date of screening visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Period from the date of the drug administration to the patient's death

OTHER OUTCOMES:
Pharmacokinetic parameters - Cmax | From date of screening visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Maximum concentration of drug by dose level
Pharmacokinetic parameters - Cmin | From date of screening visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Minimum concentration of drug by dose level
Pharmacokinetic parameters - AUC0-t | From date of screening visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Area under the curve from baseline to each timepoint by dose level
Pharmacokinetic parameters - Tmax | From date of screening visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Time of Cmax by dose level
Pharmacokinetic parameters - CL | FFrom date of screening visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Clearance by dose level
Pharmacokinetic parameters - Vd | From date of screening visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Volume of distribution by dose level
Pharmacokinetic parameters - Ke | From date of screening visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Elimination rate constant by dose level
Pharmacokinetic parameters - T½ | From date of screening visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Half-life by dose level
Change in concentration of serum angiogenic factor or receptor | From date of screening visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  VEGF, placental growth factor [PLGF], soluble vascular endothelial growth factor receptor [sVEGFR]-2, sVEGFR-1, etc.
PD-L1, VEGFR-2 expression level | From date of screening visit until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  PD-L1, VEGFR-2 expression level in tumour environment such as tumour, tumour vessel and parenchymal tissue

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Liverpool Hospital, Liverpool, New South Wales
  - Hollywood Private Hospital, Nedlands, Western Australia